CLINICAL TRIAL: NCT02260843
Title: Efficacy of Tai Chi Training to Alleviate Insomnia in Older Adults: A Randomized Controlled Trial
Brief Title: Efficacy of Tai Chi Training on Insomnia in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Angus Yu (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government); The University of Hong Kong (Other); Chinese University of Hong Kong (Other)
Responsible Party: Sponsor-Investigator, Angus Yu, Research Assistant, The Hong Kong Polytechnic University
Organization: The Hong Kong Polytechnic University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TaiChi and Insonmia
Record Dates: First submitted 2014-06-11; First posted 2014-10-09 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Insomnia; Poor Sleeping Quality
Keywords: Insomnia; Sleeping; Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Subjects in this group do not received any intervention.
- Tai Chi Intervention (Active Comparator): Subjects in this group will receive three tai chi lessons in a week while each session last for 1 hour for 12 weeks
  Interventions: Other: Tai Chi Intervention
- Generic Fitness Intervention (Placebo Comparator): Subjects in this group will receive three fitness lessons in a week while each session last for 1 hour for 12 weeks
  Interventions: Other: Generic Fitness

INTERVENTIONS:
Other: Generic Fitness — Subjects in this group will receive three fitness lessons in a week while each session last for 1 hour for 12 weeks
  Arms: Generic Fitness Intervention
Other: Tai Chi Intervention — Subjects in this group will receive three tai chi lessons in a week while each session last for 1 hour for 12 weeks
  Arms: Tai Chi Intervention

SUMMARY:
Elderly insomnia is a serious public health problem. Current conventional approaches for treating insomnia are not suitable or effective in elderly population. It has been previously demonstrated that Tai Chi has definite advantages to be developed as self-help therapy in older adults and has been preliminarily demonstrated to improve sleep in older people. This project aims to evaluate the efficacy of Tai Chi training on alleviating chronic insomnia in older adults.

DETAILED DESCRIPTION:
Elderly insomnia is a serious public health problem. It has been estimated over 50% of elderly have sustained sleep complaints. About 20-40% of the elderly worldwide are reported insomniac. In Hong Kong, a high proportion (38%) of older people have been reported to have sleep disorders. These figures are alarming because insomnia associates with co-morbidities including cognitive impairment, depression, mood/anxiety disorders, risks for falls, hypertension, and heart disease in elderly. It also destructively affects daily functioning by impairing the memory and reducing the attention span and response time. Most importantly, insomnia has been evidently shown to link with the increased risk of hospitalization and mortality. As the proportion of geriatric population is rapidly increasing, it is foreseeable that the socioeconomic impact of elderly insomnia to the healthcare system will be undoubtedly aggravated.

Current conventional approaches for treating insomnia are not suitable or effective in elderly population. Pharmacologic treatment has always been a concern in insomniac senior patients due to the adverse drug effects including dependence, abuse, cognitive impairment and increase in risk of falls and hip fractures. With fewer adverse effects and consistent efficacy, cognitive behavioral therapy (CBT) is taken as a more appropriate remedy for elderly insomnia. However, the operation of effective CBT for insomnia is very labor demanding and cost-ineffective. The large-scale use of CBT for elderly insomnia is not feasible due to the shortage of CBT specialty-trained healthcare providers and the high treatment cost. The limited availability of CBT treatment is far insufficient to match with the increasingly large demand of insomniac elderly. There is another problem with the conventional approaches. It is observed that most of the insomnia sufferers would not seek timely clinical consultation and they tend to initiate self-help treatments when facing the problem of insomnia. This situation is suggested to be more common in Chinese elderly due to the traditional Confucius philosophy of reservation and quietness probably drive them more likely to keep the problem to themselves and become reluctant to seek prompt clinical help until serious medical symptom occurs. Given the prevalence of elderly insomnia is already high and keeps increasing, there is an urgent need to explore other effective therapeutic modalities preferably in forms of self-help remedies that can help to relieve the problem of elderly insomnia.

Tai Chi has definite advantages to be developed as self-help therapy in older adults. Tai Chi, a traditional form of Chinese fitness exercise, is a unique form of physical activity of low impact and slow body movement, which includes a meditation component. It is a moderate type of exercise that is well perceived to be suitable for regular practice by older population. It is expected that Tai Chi is more acceptable to the elderly patients to be incorporated with their daily life as an instant approach for remedying insomnia relative to the conventional clinical treatment such as CBT. Additional advantages of Tai Chi include low-cost and can be conveniently practiced at any time and any place without requirement for extensive facilities. Certainly, the practice of Tai Chi is more accessible than the conventional CBT treatment, which facilitates the large-scale use of Tai Chi to relieve insomnia in elderly population. Furthermore, Tai Chi can be practiced individually or in a group. If practicing in a group, Tai Chi provides additional benefit by serving as a vehicle for establishing social interaction through which older people can establish friendship and gain supports from other seniors.

Tai Chi has a number of beneficial effects on geriatric health and fitness. These health benefits include improvements of aerobic fitness, energy metabolism, muscular strength and balance. In addition to the improvements of cardiorespiratory function, bone loss, posture stability and flexibility, Tai Chi exercise has also been shown to improve psychological well-being via relieving symptoms of anxiety and depression and reducing mood disturbances. All these physical and psychological advantages of Tai Chi cooperatively support its prescription to the senior population.

Tai Chi has been preliminarily demonstrated to improve sleep in older people. Favorable effects on sleep parameters have been reported in geriatric following 12 weeks to 6 months of Tai Chi training. The self-reported sleep quality is demonstrated to be improved by a 12-week of Tai Chi intervention in the senior residents in elderly home. Favorable effects of 12-week of Tai Chi training in patients with chronic heart failure are reported by showing the enhancement of sleep stability as assessed by sleep spectrogram. A longer period (6-month) of Tai Chi training has also been shown to improve the Pittsburgh Sleep Quality Index (PSQI)-indicated sleep quality in community-dwelling older adults. In older subjects with moderate sleep complaint or sleep-disturbance, 24/25-week of Tai Chi training is shown to improve the self-rated sleep quality, habitual sleep efficiency, sleep duration, and sleep disturbance.

All these preliminary data collectively indicate the beneficial effects of Tai Chi on improving sleep in geriatric population. Nonetheless, all these studies have a common design limitation, which is the lack of direct objective sleep measures. With the study limitation and research gaps, the present project is proposed to examine the therapeutic effects of Tai Chi on chronic insomnia in elderly by including objective sleep measures. The findings of this project are expected to have impact to unveil the efficacy of Tai Chi to alleviate elderly insomnia, which has been an epidemic healthcare problem that necessitates to be tackled promptly.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older
* ethnic Chinese
* fulfill the DSM-V criteria for chronic insomnia including difficulties to initiate sleep, maintain sleep or non-restorative sleep with complaint of impairment of daytime functioning, sleep difficulty occurs at least 3 nights per week and is present for at least three months.

Exclusion Criteria:

* cannot walk without assistive tool (e.g., cane)
* any serious somatic condition that prevent participation for Tai Chi/generic fitness activities
* current regular practicing of moderate exercise training or Tai Chi (>3 times a week of >30-min per session)
* any serious chronic diseases known to affect sleep (e.g., cancer and autoimmune diseases)
* under treatment of serious diseases known to affect sleep (e.g., cancer chemotherapy)
* any chronic pain disorders known to affect sleep.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Actigraphy-measured sleep onset latency | Immediately after completion of the 12 weeks intervention
  Objectively measured sleep onset latency (min)
Actigraphy-measured sleep efficiency | Immediately after completion of the 12 weeks intervention
  Objectively measured sleep efficiency (%)
Actigraphy-measured wake time after sleep onset | Immediately after completion of the 12 weeks intervention
  Objectively measured wake time after sleep onset (min)
Actigraphy-measured total sleep time | Immediately after completion of the 12 weeks intervention
  Objectively measured total sleep time (min)
Actigraphy-measured number of awakening | Immediately after completion of the 12 weeks intervention
  Objectively measured number of awakening (number of times) after sleep onset
Actigraphy-measured average wake time | Immediately after completion of the 12 weeks intervention
  Objectively measured average wake time (min) of all awaken time after sleep onset
Actigraphy-measured sleep onset latency | 24 months after the completion of intervention
  Objectively measured sleep onset latency (min)
Actigraphy-measured Sleep efficiency | 24 months after the completion of intervention
  Objectively measured sleep efficiency (%)
Actigraphy-measured wake time after sleep onset | 24 months after the completion of intervention
  Objectively measured wake time after sleep onset (min)
Actigraphy-measured total sleep time | 24 months after the completion of intervention
  Objectively measured total sleep time (min)
Actigraphy-measured number of awakening | 24 months after the completion of intervention
  Objectively measured number of awakening (number of times) after sleep onset
Actigraphy-measured average wake time | 24 months after the completion of intervention
  Objectively measured average wake time (min) of all awaken time after sleep onset

SECONDARY OUTCOMES:
Score of Pittsburgh Sleep Quality Index | Immediately after completion of the 12 weeks intervention and 24 months after the completion of intervention
  Pittsburgh Sleep Quality Index is a questionnaire that assess sleeping quality with scale ranged from 0 to 21. (A smaller score suggests a better sleep quality)
Change in dose of Sleep Medication | Immediately after completion of the 12 weeks intervention and 24 months after the completion of intervention
  The change in dose of sleep medication used by the subjects after intervention.
Score of Insomnia Severity Index | Immediately after completion of the 12 weeks intervention and 24 months after the completion of intervention
  Insomnia Severity Index is a questionnaire that assess sleeping quality with scale ranged from 0 to 28. (A smaller score suggests a better sleep quality)
7-day Sleep Diary | Immediately after completion of the 12 weeks intervention and 24 months after the completion of intervention
  Self-recorded sleep parameters (sleep onset latency, sleep efficiency, total sleep time, wake time after sleep onset, number of awakening and average awaken time)
Treatment response rate | Immediately after completion of the 12 weeks intervention and 24 months after the completion of intervention
  The percentage of participants that have their Score of Pittsburgh Sleep Quality Index reduced by at least 5 points
Remission rate of insomnia | Immediately after completion of the 12-week intervention and 24-month after the complete completion of the 12-week intervention
  The percentage of participants that reached to remission of chronic insomnia according to DSM-5Immediately after the completion of the 12-week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Parco MF Siu, PHD, Principal Investigator — The Hong Kong Polytechnic University
Locations (3):
- China (3):
  - The Chinese University of Hong Kong, Hong Kong, Hong Kong
  - The University of Hong Kong, Hong Kong, Hong Kong
  - The Hong Kong Polytechnic University, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices), as well as the study protocol and the statistical analysis plan, will be shared, beginning 3 months and ending 5 years following publication of the Article. Data will be shared with researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. Proposals should be directed to pmsiu@hku.hk to gain access, and data requestors will need to sign a data-access agreement.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following publication of the Article
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal to achieve aims in the approved proposal. Proposals should be directed to pmsiu@hku.hk to gain access, and data requestors will need to sign a data-access agreement.

REFERENCES:
- [Derived] Siu PM, Yu AP, Tam BT, Chin EC, Yu DS, Chung KF, Hui SS, Woo J, Fong DY, Lee PH, Wei GX, Irwin MR. Effects of Tai Chi or Exercise on Sleep in Older Adults With Insomnia: A Randomized Clinical Trial. JAMA Netw Open. 2021 Feb 1;4(2):e2037199. doi: 10.1001/jamanetworkopen.2020.37199. PMID 33587135